# Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory Biomarkers in Osteoarthritis Genu

#### **EXPLANATION SHEET TO PROSPECTIVE SUBJECTS**

We, the research team consisting of Srinalesti Mahanani, Nyoman Kertia, Desi Natalia Trijayanti Idris, Erlin Kurnia, chaired by Srinalesti Mahanani from will conducted research entitled Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory Biomarkers in Osteoarthritis Genu.

This research aims to determine the effect of a combination of turmeric extract standardized curcuminoids on secretion of TNF-Alpha, C-Reactive Protein, Interleukin-1 and Pain elderly with genu osteoarthritis.

The research team invites fathers/mothers/relatives to take part in this research. This research requires around 72 research subjects, with a period of participation each subject approximately 4 weeks - 2 months.

### A. Volunteering to participate in research

You are free to choose to participate in this research without any coercion. if you If you have decided to join, you are also free to withdraw/change mind at any time without being subject to any fines or sanctions. If you are not willing to participate then you will still get treatment at GBI Ngadinegaran in accordance with applicable procedures

#### **B. Research Procedures**

If you are willing to participate in this research, you will be asked to sign This consent form is in two copies, one for you to keep, and one for you researcher. The next procedure is:

- 1. Mr/Mrs/Br will be interviewed by a doctor to ask: Name, age, history disease, history of drug use, history of allergies, smoking habits.
- Mr/Mrs/Sdr will also be interviewed with several questions according to the questionnaire which exists. This interview aims to measure levels of anxiety and health your mentality.

Date: 20/07/2025

Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory

Biomarkers in Osteoarthritis Genu


- Mr/Mrs/Sdr will undergo a physical examination by a doctor to check the status health
- 4. Mr/Mrs/Br will undergo an X-ray examination of the knee
- If you use painkillers, you will be asked to Stop consuming for 1 week
- 6. One week later the research will begin. You will be asked to come together at the posyandu at 6.45 for further blood collection.
- 7. Blood sampling was carried out twice during the research period how to place a butterfly needle in a vein in the forearm.
  Blood collection is carried out using a butterfly needle that has been installed.
  The first collection is carried out before therapy is given in approximately one amount tablespoon, and the next intake is after the therapy is given about one tablespoon
- 8. This first blood draw is for laboratory examination regarding the condition blood and body hormones.
- 9. Blood collection is carried out by nurses who are accustomed to taking blood.
- 10. Because in this research there will be 2 groups, namely the group that given medication and therapy as well as groups who did not receive medication and therapy then Mr/Ms/Sdr will be divided into 2 groups randomly so that there are It is possible that the capsule given to you may not contain it medicinal ingredients. Respondents and researchers do not know which group they fall into, only only the therapist knows.
- 11. On the appointed day and for the next 21 days, Mr/Mrs/Br will be given

  The medicine is in capsule form which must be taken with water 3 times
  a day. And also Mr/Ms/Sdr will get a visit schedule for therapy
  acupressure. Mr/Ms/Sdr will be asked to come to the therapist's house according to the schedule.
- 12. This research will involve families to accompany respondents during the process research (the family will accompany the respondent in drinking herbal therapy, filling observation sheet for taking medication and accompanying when administering acupressure therapy as well report to researchers if unbearable pain occurs during the period study).
- 13. Researchers will involve posyandu cadres to alert patients and families taking medication and doing therapy, as well as researchers will create a system reminder to remind the family.

Date: 20/07/2025

Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory

Biomarkers in Osteoarthritis Genu


C. Obligations of research subjects

As research subjects, you are obliged to follow the rules or regulations

research instructions as written above. If something is not clear,

You can ask the researchers further questions. During the research, no

permitted to take other medicines or herbal medicines other than those given by the researcher.

D. Risks and Side Effects and Their Management

Turmeric herbal therapy interventions and acupressure massage do not provide any side effects

straight to you. During the research, researchers set up protective measures

necessary if something undesirable happens. Protection provided

by researchers is examination by a doctor and treatment in hospital.

E. Benefits

The direct benefit you get is that you get non-therapy

pharmacological to treat pain and discomfort due to Osteoarthritis Genu as well

useful for further treatment at home.

F. Confidentiality

All information relating to the identity of research subjects will be kept confidential

and will only be known to researchers, research staff and auditors. The research results will be

published without the identity of the research subjects.

**G.** Compensation

You will receive an X-ray examination to determine the condition

knee joint and will receive therapy in accordance with the provisions of the study.

Mr/Ms/Sdr will get tools for massage therapy (towel and oil).

the next will be yours. After the research activities are completed, Mr./Ms./Br

Those in the control group will receive herbal therapy and therapy

acupressure according to that received by the treatment group.

H. Financing

All costs related to research will be borne by the researcher.

Date: 20/07/2025

Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory

Biomarkers in Osteoarthritis Genu


## I. Additional Information

You are given the opportunity to ask anything that is not clear in connection with this research. If at any time side effects occur or If you need further explanation, you can contact Srinalesti Mahanani at No. Mobile phone. 085729006547.

You can also ask the Ethics Committee about research

Medical and Health Research, Faculty of Medicine, UGM (Tel. 0274-588688,
ext 17225 or +62811-2666-869; email: mhrec\_fmugm@ugm.ac.id).

Date: 20/07/2025

Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory

Biomarkers in Osteoarthritis Genu


# Efficacy Test of Curcuminoid Standardized Turmeric Capsules to Improving Inflammatory Biomarkers in Osteoarthritis Genu

## **CONSENT TO PARTICIPATE IN RESEARCH**

All these explanations have been conveyed to me and all my questions have been answered answered by the researcher. I understand that if I need an explanation, I can asked Srinalesti Mahanani.

Patient/subject signature:

(Clear name .......)

Witness signature:

(Clear name .......)